CLINICAL TRIAL: NCT00275392
Title: Vestibular Rehabilitation and Dizziness in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C4168-P
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Dizziness
Keywords: Dizziness; Geriatrics; Rehabilitation; Vestibular rehabilitation
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vestibular Rehabilitation (Experimental): vestibular exercises plus standard balance and gait exercises
  Interventions: Behavioral: Vestibular rehabilitation
- Placebo (Placebo Comparator): placebo exercises plus standard balance and gait exercises
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Vestibular rehabilitation — vestibular adaptation and substitution exercises
  Arms: Vestibular Rehabilitation
Behavioral: Placebo — placebo vestibular exercises
  Arms: Placebo

SUMMARY:
The purpose of this study is to develop effective exercise intervention to reduce dizziness and fall risk in older adults with non-specific dizziness. We hypothesize that the use of vestibular exercises can reduce dizziness and improve gaze and postural stability in older persons.

DETAILED DESCRIPTION:
Community dwelling older individuals who present to a specialty dizziness clinic (Atlanta VAMC or Emory University) with a primary complaint of dizziness will be recruited to participate in this study. Before beginning the study, the presence of normal vestibular function will be measured directly using standard vestibular function tests. Individuals will be randomly assigned to the vestibular exercise group (VR) or to the control group (CON). Data will be collected prior to the initiation of physical therapy and at the completion of the 6-week intervention period.

The VR group will perform vestibular exercises plus balance and gait exercises. The CON group will perform saccadic eye movements without targets against a blank wall, as well as balance and gait exercises. The balance and gait exercises for each group will be based on identified impairments and functional limitations, as is the standard of care in physical therapy. All subjects within a group will follow the same exercise progression for the vestibular or eye movement exercises. Subjects will be seen in the clinic on a weekly basis to review and modify the exercises according to a standard protocol and to reinforce compliance.

ELIGIBILITY:
Inclusion Criteria:

Patients must be at least 60 years of age, seeking medical care due to dizziness and have normal vestibular function based on results of the clinical examination, rotary chair and/or caloric tests.

Exclusion Criteria:

Abnormal vestibular function based on results of clinical examination, rotary chair and/or caloric tests.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D. Hall, PhD PT, Principal Investigator — Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia, United States

REFERENCES:
- [Result] Hall CD, Heusel-Gillig L, Tusa RJ, Herdman SJ. Efficacy of gaze stability exercises in older adults with dizziness. J Neurol Phys Ther. 2010 Jun;34(2):64-9. doi: 10.1097/NPT.0b013e3181dde6d8. PMID 20588090

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo exercises plus standard balance and gait exercises
  Placebo Vestibular rehabilitation: placebo vestibular exercises
Period: Overall Study
Arm/Group | Vestibular Rehabilitation | Placebo
Started | 20 | 19
Completed | 20 | 17
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vestibular Rehabilitation | Placebo | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (6.5) | 74.5 (8.5) | 73.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 3 | 6 | 9
Dynamic Gait Index [Mean (Standard Deviation); unit: units on a scale] — The Dynamic Gait Index (DGI) measures the ability to adapt gait to external demands and also is used to assess fall risk while walking. The eight items of the DGI include walking while changing speed and turning the head, walking over and around obstacles, and stair climbing. Scoring of the DGI is based on a 4-point scale from 0 to 3 with 0 indicating severe impairment and 3 indicating normal ability. A maximum total score of 24 is possible and scores of < 20 indicate risk for falling.
  units on a scale | 14.2 (3.1) | 16.1 (2.6) | 15.1 (3.0)
Dynamic Visual Acuity [Mean (Standard Deviation); unit: LogMAR] — Visual acuity during head movement (dynamic visual acuity, DVA) was measured using customized computerized software. Participants identified letters while turning the head from side to side between 120 and 180 deg/s. DVA, the difference in acuity between head stationary and moving, is reported as the average of rightward and leftward scores; higher scores indicate worse visual acuity (0.00 LogMAR = 20/20).
  LogMAR | 0.20 (0.08) | 0.14 (0.07) | 0.16 (0.08)

OUTCOME MEASURES:

1. Primary Outcome: Dynamic Gait Index
Description: Fall risk was determined using the Dynamic Gait Index (DGI). A maximum total score of 24 is possible and a total score of < 20 indicates risk for falling.
Time Frame: 6 weeks
Population: Per-protocol analyses (i.e., only subjects who completed the intervention were included).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vestibular Rehabilitation | Placebo
Number analyzed (Participants) | 20 | 17
units on a scale
  Discharge (6 weeks) | 18.9 (1.8) | 18.9 (3.0)
  Baseline | 14.2 (3.1) | 16.1 (2.6)
Statistical Analysis 1: Comparison: Vestibular Rehabilitation vs Placebo; Test type: Superiority or Other; p = 0.026, RM ANOVA — Interaction effect
Statistical Analysis 2: Comparison: Vestibular Rehabilitation vs Placebo; Test type: Superiority or Other; p < .001, RM ANOVA — main effect of time
Statistical Analysis 3: Comparison: Vestibular Rehabilitation vs Placebo; Test type: Superiority or Other; p > .05, RM ANOVA — main effect of group

2. Secondary Outcome: Dynamic Visual Acuity
Description: Visual acuity during head movement (dynamic visual acuity, DVA) was measured using customized computerized software. DVA is measured in Logarithm of the Minimum Angle of Resolution (LogMAR). Participants identified letters while turning the head from side to side between 120 and 180 deg/s. DVA, the difference in acuity between head stationary and moving, is reported as the average of rightward and leftward scores; higher scores indicate worse visual acuity.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Vestibular Rehabilitation | Placebo
Number analyzed (Participants) | 20 | 17
LogMAR
  Discharge (6 weeks) | 0.14 (0.07) | 0.19 (0.08)
  Baseline | 0.20 (0.08) | 0.21 (0.10)
Statistical Analysis 1: Comparison: Vestibular Rehabilitation vs Placebo; Test type: Superiority or Other; p > 0.05, RM ANOVA — Interaction effect
Statistical Analysis 2: Comparison: Vestibular Rehabilitation vs Placebo; Test type: Superiority or Other; p = .016, RM ANOVA — main effect of time
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority or Other; p > .05, RM ANOVA — Main effect of Group

ADVERSE EVENTS:
Arm/Group | Vestibular Rehabilitation | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes